CLINICAL TRIAL: NCT06724978
Title: A Phase 1 Single- and Multiple-ascending-dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of S-740792 in Healthy Adult Study Participants
Brief Title: A Study of S-740792 in Healthy Adult Study Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2318VA711
Record Dates: First submitted 2024-12-06; First posted 2024-12-09 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Healthy Participants
Keywords: First-in-human; S-740792; Midazolam; Bioavailability; Food Effect
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Part 3 will be a 3-sequence, 3-period crossover study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 3 will be open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (Single Ascending Dose) (Experimental): Participants will receive S-740792 or placebo.
  Interventions: Drug: S-740792 Suspension; Drug: Placebo
- Part 2 (Multiple Ascending Dose) (Experimental): Participants will receive S-740792 or placebo, in addition to midazolam.
  Interventions: Drug: S-740792 Suspension; Drug: Midazolam; Drug: Placebo
- Part 3 (Bioavailability) (Experimental): Participants will receive S-740792 as a suspension and as a tablet.
  Interventions: Drug: S-740792 Suspension; Drug: S-740792 Tablet

INTERVENTIONS:
Drug: S-740792 Suspension — Participants will receive S-740792 as an oral suspension.
Drug: Midazolam — Participants will receive midazolam as a syrup.
  Arms: Part 2 (Multiple Ascending Dose)
Drug: Placebo — Participants will receive placebo as an oral suspension.
  Arms: Part 1 (Single Ascending Dose); Part 2 (Multiple Ascending Dose)
Drug: S-740792 Tablet — Participants will receive S-740792 as an oral tablet.
  Arms: Part 3 (Bioavailability)

SUMMARY:
This is a 3-part study of S-740792 in healthy adult participants. Part 1 (single-ascending-dose and food effect) will investigate the safety, tolerability, and pharmacokinetics (PK) of S-740792. Part 2 (multiple-ascending-dose and drug-drug interaction) will investigate the safety, tolerability, and PK of S-740792, in addition, the effect of multiple doses of S-740792 on the PK of midazolam. Part 3 will investigate the relative bioavailability of S-740792 tablet compared to S-740792 suspension and the food effect on the PK of the S-740792 tablet.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index within the range 18.5 to 30.0 kilograms/meter squared (inclusive).

Key Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Participants who require medication or other treatment (for example, dietary restrictions or physical therapy).
* Participants who have participated in any other clinical study involving an investigational study intervention or any other type of medical research within 28 days or 5 half-lives of that drug (if known), whichever is longer before signing of the informed consent form for this study or who are currently participating in such a study.
* Positive test results of the following at screening or within 6 months prior to administration of study intervention:
* hepatitis B surface antigen
* hepatitis C virus antibody
* serological test for syphilis
* human immunodeficiency virus antigen/antibody
* drug screen
* alcohol screen
* Participants who have used tobacco or nicotine-containing products (including electronic-cigarette, pipe tobacco, cigar, chewing tobacco, nicotine patch, and nicotine gum) within 6 months prior to admission or a positive cotinine test at screening or on admission.

Note: Additional inclusion/exclusion criteria may apply, per protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Parts 1 and 2: Number of Participants Experiencing Treatment-emergent Adverse Events | Day 1 through Day 28
Part 3: Plasma Concentration of S-740792 | Day 1 (pre-administration, up to 144 hours post-administration) of periods 1-3 (10 days/period)
Part 3: Time to Maximum Plasma Concentration (Tmax) of S-740792 | Day 1 (pre-administration, up to 144 hours post-administration) of periods 1-3 (10 days/period)

SECONDARY OUTCOMES:
Parts 1 and 2: Plasma Concentration of S-740792 | Day 1 (pre-administration, up to 144 hours post-administration), Days 10, 14, 24, and 28
Parts 1 and 2: Time to Maximum Plasma Concentration (Tmax) of S-740792 | Day 1 (pre-administration, up to 144 hours post-administration), Days 10, 14, 24, and 28
Part 1: Plasma Concentration of S-740792 After a High-fat Meal | Day 1 (pre-administration, up to 144 hours post-administration), Day 10, and Day 14
Part 1: Tmax of S-740792 After a High-fat Meal | Day 1 (pre-administration, up to 144 hours post-administration), Day 10, and Day 14
Part 2: Plasma Concentration of Midazolam After Administration of S-740792 | Day -1 (pre-administration of midazolam) and Day 14 (up to 24 hours post-administration)
Part 2: Tmax of Midazolam After Administration of S-740792 | Day -1 (pre-administration of midazolam) and Day 14 (up to 24 hours post-administration)
Part 3: Number of Participants Experiencing Treatment-emergent Adverse Events | Day 1 through Day 62

CONTACTS AND LOCATIONS:
Locations (1):
- Fortrea Clinical Research Unit, Inc., Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No